CLINICAL TRIAL: NCT00143156
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Trial of Pregabalin Versus Placebo in the Treatment of Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Pregabalin vs Placebo in Treatment of Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081071
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2008-04

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin

INTERVENTIONS:
Drug: pregabalin

SUMMARY:
To evaluate the efficacy and safety of pregabalin administered twice a day compared to placebo in reducing pain in subjects with painful diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age, of any ethnic origin
* Type 1 or 2 diabetes mellitus
* Pain score greater than or equal to 4 on the 11-point numeric pain rating scale

Exclusion Criteria:

* Neurologic disorders unrelated to diabetic neuropathy that may confuse or confound the assessment of neuropathic pain.
* Presence of severe pain associated with conditions other than diabetic peripheral neuropathy, that could confound the assessment or self-evaluation of pain due to DPN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2005-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is the endpoint End of Week 12 weekly mean pain score derived from the pain diary.

SECONDARY OUTCOMES:
End of Week 12 responder rates, Brief Pain Inventory - short form, sleep interference scores, Medical Outcome Study - Sleep Scale, Hospital Anxiety and Depression Scale, Patient Global Impression of Change, Neuropathic Pain Inventory Symptom Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- United States (47):
  - Pfizer Investigational Site, Tuscaloosa, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Los Gatos, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Englewood, New Jersey
  - Pfizer Investigational Site, Shrewsbury, New Jersey
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Frisco, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Charlottesville, Virginia
- Pfizer Investigational Site, Ponce, Puerto Rico

REFERENCES:
- [Derived] Alexander J Jr, Edwards RA, Manca L, Grugni R, Bonfanti G, Emir B, Whalen E, Watt S, Brodsky M, Parsons B. Integrating Machine Learning With Microsimulation to Classify Hypothetical, Novel Patients for Predicting Pregabalin Treatment Response Based on Observational and Randomized Data in Patients With Painful Diabetic Peripheral Neuropathy. Pragmat Obs Res. 2019 Oct 31;10:67-76. doi: 10.2147/POR.S214412. eCollection 2019. PMID 31802967
- [Derived] Alexander J Jr, Edwards RA, Brodsky M, Manca L, Grugni R, Savoldelli A, Bonfanti G, Emir B, Whalen E, Watt S, Parsons B. Using time series analysis approaches for improved prediction of pain outcomes in subgroups of patients with painful diabetic peripheral neuropathy. PLoS One. 2018 Dec 6;13(12):e0207120. doi: 10.1371/journal.pone.0207120. eCollection 2018. PMID 30521533
- [Derived] Edwards RA, Bonfanti G, Grugni R, Manca L, Parsons B, Alexander J. Predicting Responses to Pregabalin for Painful Diabetic Peripheral Neuropathy Based on Trajectory-Focused Patient Profiles Derived from the First 4 Weeks of Treatment. Adv Ther. 2018 Oct;35(10):1585-1597. doi: 10.1007/s12325-018-0780-3. Epub 2018 Sep 11. PMID 30206821
- [Derived] Parsons B, Li C, Emir B, Vinik AI. The efficacy of pregabalin for treating pain associated with diabetic peripheral neuropathy in subjects with type 1 or type 2 diabetes mellitus. Curr Med Res Opin. 2018 Nov;34(11):2015-2022. doi: 10.1080/03007995.2018.1509304. Epub 2018 Sep 20. PMID 30084288
- [Derived] Markman JD, Jensen TS, Semel D, Li C, Parsons B, Behar R, Sadosky AB. Effects of Pregabalin in Patients with Neuropathic Pain Previously Treated with Gabapentin: A Pooled Analysis of Parallel-Group, Randomized, Placebo-controlled Clinical Trials. Pain Pract. 2017 Jul;17(6):718-728. doi: 10.1111/papr.12516. Epub 2016 Dec 1. PMID 27611736
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081071&StudyName=Pregabalin%20vs%20Placebo%20in%20Treatment%20of%20Neuropathic%20Pain%20Associated%20with%20Diabetic%20Peripheral%20Neuropathy%20